CLINICAL TRIAL: NCT02338648
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled Evaluation of the Safety and Efficacy of SUN 131 Transdermal System (TDS) as Compared to Placebo TDS in Adult Patients With a Chalazion
Brief Title: Safety and Efficacy Study of SUN 131 TDS as Compared to Placebo TDS in Adult Patients With a Chalazion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Senju USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUN-131-02
Record Dates: First submitted 2014-10-31; First posted 2015-01-14 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-06

CONDITIONS: Chalazion
MeSH Terms: conditions — Chalazion | interventions — tyramine-deoxysorbitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUN-131 1.5% TDS (Experimental): Subjects will be randomly assigned to receive SUN-131 1.5% TDS for the affected eye. All patches will be worn for 16±4 hours each day for 21 days.
  Interventions: Drug: SUN-131 1.5% TDS
- Placebo TDS (Placebo Comparator): Placebo Patch for Blinding Purposes
  Interventions: Drug: Placebo TDS

INTERVENTIONS:
Drug: SUN-131 1.5% TDS — Active transdermal patch
  Arms: SUN-131 1.5% TDS
Drug: Placebo TDS — Placebo transdermal patch for blinding
  Arms: Placebo TDS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SUN-131 1.5% TDS as compared with placebo TDS in the treatment of chalazion based on the proportion of subjects that have complete response. Complete response is defined as the absence of any significant clinical signs of a chalazion with possible scaring or skin defects resulting from healing of the chalazion allowed.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to receive one of the following treatments in the affected eyelid:

* SUN-131 1.5% TDS (n=30)
* Placebo TDS (n=30)

At baseline prior to application of the TDS an assessment will be performed on both the subject's eyes including the chalazion site itself.

All subjects will return to the site on Days 8±1, 15±2 and 23±2 for evaluations. During the the 23±2 visit, a clinical evaluation will be performed to determine if the chalazion is still present.

There will also be follow up on Day 29±3, and on Day 50 visit (study days 47 to 60) to evaluate the safety and durability of the effect of the SUN-131 1.5% TDS.

Data review and safety assessments will be conducted by the medical monitor periodically throughout the trial and at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older of either sex and any race
* Chalazion with visible single granuloma in an upper or lower eyelid. If more than one eyelid is diagnosed with a chalazion, the most inflammatory chalazion shall be selected as the study eyelid. Other eyelids containing a chalazion will not be treated with investigational product in this trial.
* Chalazion intended for study treatment presents no more than 3 weeks based on subject history.
* Normal lid function
* Must be willing and able to correctly apply and wear a transdermal patch to the eyelid for 16±4 hours each day for repeated application
* Female subjects of childbearing potential must have a negative urine pregnancy test on Day 1, and must agree to use method of contraception from the start of study drug use and for 30 days after discontinuation of study drug. Approved methods of contraception include, an IUD with spermicide, a female condom with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, use of a condom with spermicide by sexual partner or a sterile sexual partner or oral contraceptives.
* If male, subjects must be sterile or willing to use an approved method of contraception from the time of study drug administration to 30 days after discontinuation of study drug. Males must be willing to refrain from sperm donation within 30 days after study drug treatment.
* Are able and willing to attend all study visits and follow all study instructions.
* Have signed written informed consent before undergoing any study related procedures and is willing to comply with all study procedures.
* Avoid wearing contact lenses or any new facial cosmetic products during the study trial period.

Exclusion Criteria:

* Chalazion which have atypical features (a recurring chalazion at the same spot, abnormal surrounding lid tissue, associated loss of tissues).
* Chalazion at the lid margin.
* Active ocular or eyelid infection (bacterial, viral, or fungal), any ocular or eyelid condition that in the investigator's opinion could affect the subject's health or the study parameters.
* An abnormal skin condition on the upper and lower eyelid region of the eyelid (e.g. eczema, psoriasis, etc.) where the patches will be applied.
* Intraocular pressure greater than 22 mmHg.
* Diagnosed with glaucoma.
* Use of oral and ocular therapy with a steroid within 7 days prior to administration of the study medication and during the study.
* Female subjects who are pregnant or lactating.
* Known allergy or sensitization to the test article or any formulation components.
* Major non-ocular surgery within 30 days prior to Day 1.
* History or evidence of ocular surgery within the past 3 months and/or a history of refractive surgery within the past 6 months.
* Planned surgery (ocular or systemic) during the trial period or within 30 days of removal of the transdermal patch.
* Participation in an investigational study within 30 days prior to Day 1.
* Have any ocular condition that requires chronic use of topical ophthalmic medication (e.g., glaucoma, dry eye, allergic conjunctivitis) with exception of artificial tear drops or lubricant eye drops or that, in the investigator's opinion, prevents the safe use of the patch.
* History of any previous functional or cosmetic eyelid surgery (including blepharopigmentation).
* Any other condition that, in the opinion of the investigator, renders the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Complete Response | Day 23±2
  Complete response is defined as the absence of any significant clinical signs of a chalazion with possible scaring or skin defects resulting from healing of the chalazion allowed.

SECONDARY OUTCOMES:
Change in Chalazion Size | Study days 47 to 60
  Size of the chalazion will be assessed using a caliper and measured as height and width in mm.
Change in Chalazion Erythema | Study days 47 to 60
  Erythema of the chalazion site itself will be assessed using a 5-point scale (i.e. 0 = no signs of erythema; to 4 = severe erythema)
Pain Associated with the Chalazion | Study days 47 to 60
  Pain assessments will be done at the clinical site using a 100 mm visual analog scale.
Time to Complete Response of the Target Chalazion | Study days 47 to 60
Durability of Response | Study days 47 to 60
  Clinical assessment of the presence of a chalazion if there was a complete response by Day 23±2.
Comparison of Adverse Event Rates and Skin Irritation between Treatment Arms | Day 23±2

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - WCCT Global Ophthalmology Research, Santa Ana, California
  - Corneal Consultants of Colorado, P.C., Littleton, Colorado
  - George Washington University Medical Faculty Association, Washington D.C., District of Columbia
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cornerstone Eye Care, High Point, North Carolina
  - Virginia Eye Consultants, Norfolk, Virginia

REFERENCES:
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Draize JH. Dermal toxicity. Appraisal of Chemicals in Food, Drugs and Cosmetics: The Association of Food and Drug Officials of the United States (3rd printing 1975); 1959. p. 46-59
- [Result] Ho SY, Lai JS. Subcutaneous steroid injection as treatment for chalazion: prospective case series. Hong Kong Med J. 2002 Feb;8(1):18-20. PMID 11861988
- [Result] Kaimbo Wa Kaimbo D, Nkidiaka MC. [Intralesional corticosteroid injection in the treatment of chalazion]. J Fr Ophtalmol. 2004 Feb;27(2):149-53. doi: 10.1016/s0181-5512(04)96109-8. French. PMID 15029042
- [Result] Ben Simon GJ, Huang L, Nakra T, Schwarcz RM, McCann JD, Goldberg RA. Intralesional triamcinolone acetonide injection for primary and recurrent chalazia: is it really effective? Ophthalmology. 2005 May;112(5):913-7. doi: 10.1016/j.ophtha.2004.11.037. PMID 15878075
- [Result] Ben Simon GJ, Rosen N, Rosner M, Spierer A. Intralesional triamcinolone acetonide injection versus incision and curettage for primary chalazia: a prospective, randomized study. Am J Ophthalmol. 2011 Apr;151(4):714-718.e1. doi: 10.1016/j.ajo.2010.10.026. Epub 2011 Jan 22. PMID 21257145
- [Result] Elsevier BH. Clinical Ocular Pharmacology. 5th Edition ed2008.